CLINICAL TRIAL: NCT06112067
Title: Efficacy and Safety of Combo-stim Deep Brain Stimulation for Treatment-refractory Mental Disorders: a Multi-center, Single Arm, Prospective, Open-label, Extendable Study
Brief Title: Efficacy and Safety of Combo-stim Deep Brain Stimulation for Treatment-refractory Mental Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: SceneRay Corporation, Limited (Industry); Huashan Hospital (Other); Shanghai 6th People's Hospital (Other); Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhen Wang, Principal investigator, Shanghai Mental Health Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBS-TRP-01
Record Dates: First submitted 2023-10-08; First posted 2023-11-01 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Deep Brain Stimulation
Keywords: deep brain stimulation; nucleus accumbens; anterior limb of internal capsule; obsessive-compulsive disorder; schizophrenia; bipolar with depression; anorexia nervosa; gambling disorder; adult autism
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Schizophrenia; Anorexia Nervosa; Gambling; Autistic Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DBS intervention group (Experimental): This is a single arm, prospective, open label clinical study, participants who fit inclusion standards, don't fit exclusion standards and fit surgical implantation standard will start DBS system stimulation and adjust parameters after 7-14 days of implantation. Then after stimulation for 8-24 weeks, they will be evaluated for treatment efficacies. This study is extendable, with agreements from participants, long term efficacy and safety follow-up study will be performed after 24 weeks ± 7 days, specific plan depends on different mental disorders.
  Interventions: Device: deep brain stimulation

INTERVENTIONS:
Device: deep brain stimulation — DBS electrodes will be implanted into the ALIC and the NAcc, electric stimulation of those areas are used to treat mental disorders and to evaluate the efficacy and safety of DBS system.

SUMMARY:
This is a multi-center, single arm, prospective, open-label, extendable study for the efficacy and safety of combo-stim deep brain stimulation for treatment-refractory mental disorders (obsessive-compulsive disorder, schizophrenia, bipolar with depression, anorexia nervosa, gambling disorder and adult autism).

DETAILED DESCRIPTION:
Total of 18 subjects from Shanghai Mental Health Center who fit inclusion and don't fit exclusion criteria are recruited to undergo neurosurgical implantation of combo-stim DBS in bilateral nucleus accumbens (NAcc) and anterior limb of internal capsule (ALIC) on a certain date, the DBS system will be turned on for stimulation and parameters adjusted 7-14 days after implantation, treatment purposes are evaluated after system has been turned on for 8-24 weeks. Primary efficacy is evaluated by change in Yale-Brown Obsessive-Compulsive Scale (Y-BOCS), Positive and Negative Syndrome (PANSS), Montgomery-Asberg Depression Rating Scale (MADRS), Body Mass Index (BMI), Autism Behavior Checklist (AuBC) score and longest consecutive days without gambling within one month. Safety is evaluated by adverse events (AE) and device-related adverse events (ADE), serious adverse events (SAE) and serious device-related events (SADE), device deficiencies (DD) and device malfunction, physical examination and vital signs, laboratory examination, electrocardiogram (ECG), imaging examination, scale evaluation and early drop out ratio due to AE.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment refractory obsessive-compulsive disorder:

   1. Aged 18~65 when signing informed consent, outpatient or inpatient, male or female.
   2. Fits DSM-5 obsessive-compulsive disorder criteria.
   3. Fits treatment refractory obsessive-compulsive disorder criteria (both i and ii):

   i.Treated with at least 3 kinds of serotonin reuptake inhibitors (SSRIs) with at least 2 kinds of 2nd generation antipsychotic medication as enhancement, enough dosage and enough course of treatment, and still no effect or intolerant.

   ii.While using enough dosage of SSRIs, treated with more than 8~12 times of Cognitive Behavior Therapy (CBT) or CBT-intolerant.

   d)Y-BOCS score ≥ 25 in screening period and baseline. e)CGI-S score ≥ 4 in screening period and baseline. f)Patient and guardian agree to DBS implant and sign informed consent after fully understood research aims, contents, anticipated treatments and risks.
2. Treatment refractory schizophrenia:

   1. Aged 18~65 when signing informed consent, outpatient or inpatient, male or female.
   2. Fits DSM-5 schizophrenia criteria.
   3. Course of disorder ≥ 5 years.
   4. Fits treatment refractory schizophrenia criteria, one of the conditions below:

   i.Treated with more than 2 different anti-psychotic medications (clozapine excluded), enough dosage (equivalent dosage as chlorpromazine ≥ 600mg/day), enough course of treatment (≥ 12 weeks), no effect or intolerant.

   ii.Treated with enough dosage of clozapine (≥ 300mg/day or blood medication concentration ≥ 350ng/ml, enough course of treatment (≥ 12 weeks), no effect or intolerant.

   e)PANSS score ≥ 70 in screening period and baseline, and at least 1 item from 5 items (P1, P2, P3, P5, P6) of PANSS positive symptom scale ≥ 4; or at least 3 items from PANSS negative symptom scale (N1~N7) ≥ 4, or at least 2 items ≥ 5.

   f)CGI-S ≥ 4 in screening period and baseline. g)GAF ≤ 60 in screening period and baseline. h)Patient and guardian agree to DBS implant and sign informed consent after fully understood research aims, contents, anticipated treatments and risks.
3. Treatment refractory bipolar with depression:

   1. Aged 18~65 when signing informed consent, outpatient or inpatient, male or female.
   2. Fits DSM-5 bipolar I or bipolar II criteria, currently with depression episode.
   3. Course of disorder ≥ 2 years.
   4. Fits treatment refractory bipolar with depression criteria (treated with two different kinds of treatment below, enough dosage and enough course of treatment ≥ 8 weeks, and cannot acquire symptom cure for 8 consecutive weeks, either i or ii):

   i.Used at least two medications (alone) among Olanzapine (10-20mg/d) + Fluoxetine (20-60mg/d), Quetiapine (200-600mg/d), Lurasidone (40-160mg/d), Lamotrigine (200-400mg/d) ii.Used at least one medication above (alone), and used one of medication above with another medication among Lamotrigine (200-400mg/d), Valproate (1000-2000mg/d) and lithium salt (blood lithium reaches 0.8mmol/L).

   e)Upon medication treatment, electroconvulsive therapy ≥ 12 times, no effect or failed (such as intolerant).

   f)Fits severe symptom criteria: i.Depression episode ≥ 12 weeks in screening period. ii.MADRS score ≥ 26 in screening period and baseline. iii.GCI-BP score ≥ 4 in screening period and baseline. iv.YMRS score ≥ 12 in screening period and baseline. g)Patient and guardian agree to DBS implant and sign informed consent after fully understood research aims, contents, anticipated treatments and risks.
4. Treatment refractory anorexia nervosa:

   1. Aged 18~65 when signing informed consent, outpatient or inpatient, male or female.
   2. Fits DSM-5 anorexia nervosa criteria, consider both restricting type and binge-eating/purging type.
   3. 10 ≤ BMI < 16 in screening period and baseline.
   4. Fits treatment refractory anorexia nervosa criteria (both i, ii, iii and iv):

   i.Course of disorder ≥ 5 years, severe and sustained anorexia nervosa. ii.With ≥ 3 times repeated inpatient history and bad treatment effect (can't complete treatment or immediate relapse after treatment).

   iii.Through systemic nutrient treatment, medication (SSRIs and/or anti-psychotics), psychotherapies (such as reinforced CBT, FBT treatment), no effect or intolerant.

   iv.Worsened instability of clinical treatment, refuse treatment or bad reaction to reinforced treatment, last for more than 1 year, with more than 2 times of involuntary food intake.

   e)Patient and guardian agree to DBS implant and sign informed consent after fully understood research aims, contents, anticipated treatments and risks.
5. Gambling disorder:

   1. Aged 18~65 when signing informed consent, outpatient or inpatient, male or female.
   2. Course of disorder ≥ 2 years.
   3. Diagnosed as gambling disorder based on DSM-5, fits medium or severe diagnostic standard (≥ 6 terms)
   4. Received systemic treatment (such as medication and social mental intervention) but still has iterative thoughts of impulse or gambling behaviors.
   5. Patient and guardian agree to DBS implant and sign informed consent after fully understood research aims, contents, anticipated treatments and risks.
6. Adult autism:

   1. Aged 18~65 when signing informed consent, outpatient or inpatient, male or female.
   2. Fits DSM-5 autism spectrum disorder diagnostic standard, and there's severe, life-threatening iterative behaviors, and independently evaluated by two psychiatric doctors.
   3. AuBC score ≥ 62 in screening period and baseline.
   4. CGI-S score ≥ 4 in screening period and baseline.
   5. Course of disorder ≥ 10 years, received systemic behavior intervention or training ( such as critical reaction training, cognitive behavior intervention, language expression training, demonstration method, natural environment training, patriarch training, social skill training, intervention based on story tales, etc. ) but failed, or intolerant.
   6. Patient and guardian agree to DBS implant and sign informed consent after fully understood research aims, contents, anticipated treatments and risks.

Exclusion Criteria:

1. With mental disorders including physical mental disorders, paranoid personality disorder, delayed mental development etc.
2. Through clinical evaluation by investigators, there exists significant suicide behavior risk.
3. From screening period to baseline, patients who has significant improvement in evaluation scores:

   1. Obsessive compulsive disorder: Y-BOCS score decreased (or improved) ≥ 20%
   2. Schizophrenia: PANSS score decreased (or improved) ≥ 20%
   3. Bipolar with depression: MADRS score decreased (or improved) ≥ 20%
   4. Anorexia nervosa: BMI improved ≥ 20%
   5. Gambling: through evaluation by investigators, online gambling behavior is significantly improved
   6. Adult autism: AuBC score decreased (or improved) ≥ 20%.
4. With severe or unstable cardiovascular, inspiratory, liver, kidney, blood, endocrine, neural system or other system disorders.
5. Has neural system disorders including physical brain disorders, brain trauma, treatment-refractory seizure etc.
6. During screening period or baseline, abnormalities in patient's physical examination, laboratory examination, electrocardiogram examination, imaging examination have significant clinical meaning, and patients who are considered unfit by investigators.
7. Implanted artificial cochlea, pacemaker, similar single-side or double-side products or experienced other physical surgeries within half a year that are considered to have effect on this trial by investigators.
8. DBS implant surgery taboos present and is considered unfit by investigators.
9. Diagnosed as HIV positive.
10. Female in gestation, lactation, or blood HCG / urine gestation test positive. Or patients who can't take effective contraception actions during the trial. Or patients planning to birth or give birth after the trial begins for 3 months.
11. Currently involved or involved in other medication or medical device clinical trials 3 months before the screening period.
12. Other patients who are considered unfit by investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
change of Y-BOCS score compared to baseline after 12 weeks of stimulation | 12 weeks.
  change of Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) score compared to baseline after 12 weeks of stimulation. The Y-BOCS is a test to rate the severity of obsessive-compulsive disorder (OCD) symptoms. Total of 10 items, total score is 40, minimum score is 0 (no symptom) , maximum score is 40 (extreme).
reduce rate of PANSS score compared to baseline after 12 weeks of stimulation | 12 weeks
  reduce rate of Positive and Negative Syndrome Scale (PANSS) score compared to baseline after 12 weeks of stimulation. The PANSS is a medical scale used for measuring symptom severity of patients with schizophrenia. Composed of three scles: The positive scale has 7 items (minimum score 7, maximum score 49), negative scale has 7 items (minimum score 7, maximum score 49), general psychopathology scale has 16 items (minimum score 16, maximum score 112). Together, PANSS total score minimum 30 (no symptom), maximum 210 (extreme).
change of Montgomery-Åsberg Depression Rating Scale (MADRS) score compared to baseline after 12 weeks of stimulation | 12 weeks
  change of Montgomery-Åsberg Depression Rating Scale (MADRS) score compared to baseline after 12 weeks of stimulation. The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Total score is 54, minimum score 0 (normal/symptom absent), maximum score 54 (severe).
change of BMI compared to baseline after 12 weeks of stimulation | 12 weeks
  change of BMI compared to baseline after 12 weeks of stimulation. Weight and height will be combined to report BMI in kg/m^2.
the duration of abstinence in gambling disorder | within 24 weeks
  within 24 weeks of stimulation, longest consecutive days without gambling
change of AuBC score compared to baseline after 12 weeks of stimulation | 12 weeks
  change of Autism Behavior Checklist (AuBC) score compared to baseline after 12 weeks of stimulation. The Autism Behavior Checklist (AuBC) is a 57-item behavior rating scale assessing the behaviors and symptoms of autism for children 3 and older. Total score 228, minimum score 57, maximum score 228.

SECONDARY OUTCOMES:
Treatment efficacy rate in OCD | within 24 weeks
  the number of treatment-response patient/total patient*100% after 8/12/24 weeks of stimulation. The Y-BOCS score reduce rate ≥ 35% and Clinical Global Impression Scale (CGI-I) score being 1 or 2 means treatment response.
Change in Y-BOCS score compared to baseline after 8/24 weeks of stimulation. Change of Y-BOCS score in OCD | within 24 weeks
  Change in Y-BOCS score compared to baseline after 8/24 weeks of stimulation. The Y-BOCS is a test to rate the severity of obsessive-compulsive symptoms. Total of 10 items, total score is 40, minimum score is 0 (no symptom) , maximum score is 40 (extreme).
Change of CGI-S score in OCD | within 24 weeks
  Change in CGI-S score compared to baseline after 8/12/24 weeks of stimulation. The clinical global impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. It is composed of Severity of Illness (CGI-S) and Global Improvement (CGI-I). Item or total score is not available for both scales, minimum score 0 (no symptom), maximum score 7 (extreme).
Change of HAMD-17 score in OCD | within 24 weeks
  Change in Hamilton Depression Scale (HAMD-17) score compared to baseline after 8/12/24 weeks of stimulation. This is a 17-item clinician-rated scale that is used to measure the severity of depression. Total score is 52, minimum socre is 0 (no symptom), maximum score is 52 (severe).
Change of HAMA score in OCD | within 24 weeks
  Change in Hamilton Anxiety Scale (HAMA) score compared to baseline after 8/12/24 weeks of stimulation. This is a psychological questionnaire used by clinicians to rate the severity of a patient's anxiety.The scale consists of 14 items, total score is 56, minimum score 0 (no symptom), maximum score 52 (severe).
CGI-I score in OCD | within 24 weeks
  CGI-I score after 8/12/24 weeks of stimulation. The clinical global impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. It is composed of Severity of Illness (CGI-S) and Global Improvement (CGI-I). In CGI-I, minimum score 1 (very much improved), maximum score 7 (extremely deteriorated).
Sheehan Disability Scale score in OCD | within 24 weeks
  Change in Sheehan Disability Scale (SDS) score compared to baseline after 8/12/24 weeks of stimulation. The Sheehan Disability Scale (SDS) is a short, simple, and cost-effective measure of disability and functional impairment. Total of 5 items, no total score/maximum/minimum score available.
Treatment efficacy rate in schizophrenia | within 24 weeks
  Treatment efficacy rate (PANSS score reduce rate ≥ 20% compared to baseline) after 8/12/24 weeks of stimulation. The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia. Composed of three scles: The positive scale has 7 items (minimum score 7, maximum score 49), negative scale has 7 items (minimum score 7, maximum score 49), general psychopathology scale has 16 items (minimum score 16, maximum score 112). Together, PANSS total score minimum 30 (no symptom), maximum 210 (extreme).
Reduce rate of PANSS score in schizophrenia | within 24 weeks
  Reduce rate of PANSS score compared to baseline after 8/24 weeks of stimulation.
Reduce rate of PANSS positive symptoms | within 24 weeks
  Reduce rate of PANSS positive symptoms compared to baseline after 8/12/24 weeks of stimulation.
Reduce rate of PANSS negative symptoms | within 24 weeks
  Reduce rate of PANSS negative symptoms compared to baseline after 8/12/24 weeks of stimulation.
Change in Global Assessment of Function (GAF) score in schizophrenia | within 24 weeks
  e)Change in Global Assessment of Function (GAF) score compared to baseline after 8/12/24 weeks of stimulation. The Global Assessment of Functioning (GAF) is a numeric scale used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of an individual. Total of 10 items, toal score 100, minimum score 1 (severely impaired), maximum score 100 (extremely high functioning).
Change of CGI-S score in schizophrenia | within 24 weeks
  Change in CGI-Schizophrenia score compared to baseline after 8/12/24 weeks of stimulation. The clinical global impression-schizophrenia (CGI-S) scale is a valid, reliable instrument to evaluate severity and treatment response in schizophrenia. Total of 5 items, total score 35, minimum score 5, maximum score 35.
CGI-I score in schizophrenia | within 24 weeks
  Change in CGI-I score compared to baseline after 8/12/24 weeks of stimulation. The clinical global impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. It is composed of Severity of Illness (CGI-S) and Global Improvement (CGI-I). In CGI-I, minimum score 1 (very much improved), maximum score 7 (extremely deteriorated).
Change of MADRS score in bipolar with depression | within 24 weeks
  Change in MADRS score compared to baseline after 8/24 weeks of stimulation. The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Total score is 54, minimum score 0 (normal/symptom absent), maximum score 54 (severe).
Treatment efficacy rate in bipolar with depression | within 24 weeks
  Treatment efficacy rate (ratio of patients whose MADRS score reduce ≥ 50% compared to baseline) after 8/12/24 weeks of stimulation. The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Total score is 54, minimum score 0 (normal/symptom absent), maximum score 54 (severe).
Symptom relieve rate in bipolar with depression | within 24 weeks
  Symptom relieve rate (ratio of patients whose MADRS score ≤ 12) after 8/12/24 weeks of stimulation. The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Total score is 54, minimum score 0 (normal/symptom absent), maximum score 54 (severe).
Change of HAMD-17 score in bipolar with depression | within 24 weeks
  Change of HAMD-17 score compared to baseline after 8/12/24 weeks of stimulation. The Hamilton Depression Rating Scale (HAMD 17) is a 17-item clinician-rated scale that is used to measure the severity of depression. Total score is 52, minimum score is 0 (no symptom), maximum score is 52 (extreme).
Change of YMRS score in bipolar with depression | within 24 weeks
  Change of Young Manic Rating Scale (YMRS) score compared to baseline after 8/12/24 weeks of stimulation. The Young Mania Rating Scale (YMRS) is an eleven-item multiple choice diagnostic questionnaire which psychiatrists use to measure the presence and severity of mania and associated symptoms. The scale has eleven items and is based on the patient's subjective report of his or her clinical condition, total score is 60, minimum score 0 (no symptom), maximum score 60 (extreme).
Change of CGI-BP-S score in bipolar with depression | within 24 weeks
  Change of CGI-BP-S score compared to baseline after 8/12/24 weeks of stimulation. The CGI-BP-S is a scale which assesses a participant's severity of their overall bipolar illness, depression, and mania. Total of 3 subscales, total score is 7 for each scale, minimum score 1, maximum score 7.
CGI-I score in bipolar with depression | within 24 weeks
  CGI-I score after 8/12/24 weeks of stimulation. The clinical global impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. It is composed of Severity of Illness (CGI-S) and Global Improvement (CGI-I). In CGI-I, minimum score 1 (very much improved), maximum score 7 (extremely deteriorated).
Change of Pittsburgh Sleep Quality Index (PSQI) in bipolar with depression | within 24 weeks
  Change of Pittsburgh Sleep Quality Index (PSQI) score compared to baseline after 8/12/24 weeks of stimulation. The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. Total of 19 items, total score 21, minimum score 0, maximum score 21.
Change of SDS in bipolar with depression | within 24 weeks
  Change of SDS score compared to baseline after 8/12/24 weeks of stimulation. The Sheehan Disability Scale (SDS) is a short, simple, and cost-effective measure of disability and functional impairment. Total of 5 items, no total score/maximum/minimum score available.
Change of BMI in anorexia nervosa | within 24 weeks
  Change of BMI compared to baseline after 8/24 weeks of stimulation. Weight and height will be combined to report BMI in kg/m^2.
Change of Eating Disorder Examination Questionnaire 6.0 in anorexia nervosa | within 24 weeks
  Change of Eating Disorder Examination Questionnaire 6.0 (EDEQ-6.0) score compared to baseline after 8/12/24 weeks of stimulation. The Eating Disorder Examination Questionnaire 6.0 (EDE-Q 6.0) is one of the most broadly used self-report tools that assesses attitudes and behaviors associated with eating disorders (EDs). Total of 28 items, there's no total score or maximum/minimum score.
Change of CGI-S score in anorexia nervosa | within 24 weeks
  Change of CGI-S score compared to baseline after 8/12/24 weeks of stimulation. The clinical global impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. It is composed of Severity of Illness (CGI-S) and Global Improvement (CGI-I). Item or total score is not available for both scales, minimum score 0 (no symptom), maximum score 7 (extreme).
Change of HAMD-17 score in anorexia nervosa | within 24 weeks
  Change of HAMD-17 score compared to baseline after 8/12/24 weeks of stimulation. The Hamilton Depression Rating Scale (HAMD 17) is a 17-item clinician-rated scale that is used to measure the severity of depression. Total score is 52, minimum score is 0 (no symptom), maximum score is 52 (extreme).
Change of HAMA score in anorexia nervosa | within 24 weeks
  Change of HAMA score compared to baseline after 8/12/24 weeks of stimulation. This is a psychological questionnaire used by clinicians to rate the severity of a patient's anxiety.The scale consists of 14 items, total score is 56, minimum score 0 (no symptom), maximum score 52 (severe).
Change of Y-BOCS score in anorexia nervosa | within 24 weeks
  Change of Y-BOCS score compared to baseline after 8/12/24 weeks of stimulation. The Y-BOCS is a test to rate the severity of obsessive-compulsive symptoms. Total of 10 items, total score is 40, minimum score is 0 (no symptom) , maximum score is 40 (extreme).
Change of Barratt Impulsivity Scale-11 in anorexia nervosa | within 24 weeks
  Change of Barratt Impulsivity Scale-11 (BIS-11) score compared to baseline after 8/12/24 weeks of stimulation. The Barratt Impulsiveness Scale (BIS) is a widely used measure of impulsiveness. Total of 26 items, there's no total score or maximum/minimum score.
CGI-I score in anorexia nervosa | within 24 weeks
  CGI-I score after 8/12/24 weeks of stimulation. The clinical global impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. It is composed of Severity of Illness (CGI-S) and Global Improvement (CGI-I). In CGI-I, minimum score 1 (very much improved), maximum score 7 (extremely deteriorated).
duration of abstinence in gambling disorder | within 24 weeks
  within 24 weeks of stimulation, total days of sustained quit gambling
Subjective craving in gambling disorder | within 24 weeks
  Change of Visual Analogue Scale (VAS) (0-10 scale, 0 is no craving, 10 is extreme craving) score compared to baseline after 8/12/24 weeks of stimulation.
Change of HAMD-17 in gambling disorder | within 24 weeks
  Change in HAMD-17 score compared to baseline after 8/12/24 weeks of stimulation. The Hamilton Depression Rating Scale (HAMD 17) is a 17-item clinician-rated scale that is used to measure the severity of depression. Total score is 52, minimum score is 0 (no symptom), maximum score is 52 (extreme).
Change of HAMA in gambling disorder | within 24 weeks
  Change in HAMA score compared to baseline after 8/12/24 weeks of stimulation. This is a psychological questionnaire used by clinicians to rate the severity of a patient's anxiety.The scale consists of 14 items, total score is 56, minimum score 0 (no symptom), maximum score 52 (severe).
Change of SDS in gambling disorder | within 24 weeks
  Change in SDS score compared to baseline after 8/12/24 weeks of stimulation. The Sheehan Disability Scale (SDS) is a short, simple, and cost-effective measure of disability and functional impairment. Total of 5 items, no total score/maximum/minimum score available.
Change of AuBC score in autism disorder | within 12 weeks
  Change in AuBC score compared to baseline after 8/24 weeks of stimulation. The Autism Behavior Checklist (AuBC) is a 57-item behavior rating scale assessing the behaviors and symptoms of autism for children 3 and older. Total score 228, minimum score 57, maximum score 228.
Change of Aberrant Behavior Checklist (AbBC) scorein autism disorder | within 24 weeks
  Change in Aberrant Behavior Checklist (AbBC) score compared to baseline after 8/12/24 weeks of stimulation. The Aberrant Behavior Checklist (AbBC) is a symptom checklist for assessing problem behaviors of children and adults with developmental disabilities. Total of 58 items, total score 174, minimum score 0, maximum score 174.
Change of GCI-S score in autism disorder | within 24 weeks
  Change in GCI-S score compared to baseline after 8/12/24 weeks of stimulation. The clinical global impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. It is composed of Severity of Illness (CGI-S) and Global Improvement (CGI-I). Item or total score is not available for both scales, minimum score 0 (no symptom), maximum score 7 (extreme).
CGI-I score in autism disorder | within 24 weeks
  CGI-I score after 8/12/24 weeks of stimulation. The clinical global impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. It is composed of Severity of Illness (CGI-S) and Global Improvement (CGI-I). In CGI-I, minimum score 1 (very much improved), maximum score 7 (extremely deteriorated).
Change of ADL score in autism disorder | within 24 weeks
  Change in Activity of Daily Living Scale (ADL) score compared to baseline after 8/12/24 weeks of stimulation. Activities of daily living (ADL) is a scale used in healthcare to refer to people's daily self-care activities. Total of 14 items, total score 56, minimum score 14, maximum score 56.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, MD,PhD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China